CLINICAL TRIAL: NCT07149207
Title: Intraoperative Molecular Imaging Using ICG for Head and Neck Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jason Newman, Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 103776
Record Dates: First submitted 2025-07-31; First posted 2025-08-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma Head and Neck Cancer (HNSCC); Margin Assessment
Keywords: Cancer; surgical margins; head and neck cancer; mucosal squamous cell cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasms; Margins of Excision | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm trial (Experimental)
  Interventions: Drug: Indocyanine Green (ICG)

INTERVENTIONS:
Drug: Indocyanine Green (ICG) — Dose: 5 mg/kg IV injection prior to surgery

SUMMARY:
This study is for adult patients with head and neck cancer who are at risk of recurrence. The purpose of this study is to evaluate whether the use of Indocyanine Green (ICG) dye allows for better identification of tumor tissue during surgical procedures. Participation will include standard of care visits along with administration of ICG dye and imaging during surgery. Participation in this study will last approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Squamous cell carcinoma of head and neck mucosal origin
* Good operative candidate
* Capable of giving informed consent

Exclusion Criteria:

* Pregnant women
* Known allergy to iodides or shellfish
* Currently incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Estimates of sensitivity and specificity using ICG. | From time of surgery until final pathology results are available (about 2 weeks)
  Sensitivity (specificity) will be estimated as the proportion of pathologically positive (negative) samples that do (do not) fluoresce using ICG.

SECONDARY OUTCOMES:
Frequency and proportion of samples for which visualization is altered using dimension. | From surgery until final pathology results are available (about 2 weeks)
  The frequency and proportion of samples for which visualization is altered (normal vs abnormal) will be summarized in each dimension (anterior, posterior, left and right lateral, superficial, deep).
Estimates of sensitivity and specificity using white light visualization. | From surgery until final pathology results are available (about 2 weeks).
  Sensitivity and specificity point and interval estimates of white light visualization relative to pathology gold standard will be constructed as described for ICG.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Newman, MD, FACS, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina, United States